CLINICAL TRIAL: NCT07332624
Title: Instant Message-delivered Acceptance and Commitment Therapy (ACT) for Neuropsychiatric Symptoms in Persons Living With Mild Cognitive Impairment: a Pilot Randomised Controlled Trial
Brief Title: Instant Message-delivered Personalised Acceptance and Commitment Therapy (ACT) for Neuropsychiatric Symptoms in Persons With Mild Cognitive Impairment
Acronym: iact
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: iact2025
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: mild cognitive impairment; acceptance and commitment therapy; neuropsychiatric symptoms
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in intervention group will receive the EMI for 8 weeks. Based on the steps of mobile message development recommended by Abroms, et al., our team will develop an ACT message content library and protocol for IM delivery (i.e. EMI).
  Interventions: Behavioral: Automated instant message-guided neuropsychiatric symptoms management
- Control group (No Intervention): The control group will receive instant messages about general mental health management from the HKSAR Government website, which is open to the public (https://www.shallwetalk.hk/en/mental-well-being/mental-well-being-is-related-to-you/), with reminder text messages of follow-up surveys.

INTERVENTIONS:
Behavioral: Automated instant message-guided neuropsychiatric symptoms management — Participants in intervention group will receive the EMI for 8 weeks. Based on the steps of mobile message development recommended by Abroms, et al., we will develop a message content library and protocol for EMI delivery.
  Arms: Intervention group

SUMMARY:
This pilot study aims to develop an automated instant message-delivered intervention (i.e., EMI) for people with mild cognitive impairment, and to investigate the feasibility and effectiveness of the intervention.

DETAILED DESCRIPTION:
1. Message contents: The message content library will consist of two parts: 1. brief mild cognitive impairment messages (optional), and 2. acceptance and commitment therapy messages (mandatory).
2. Message delivery

   * Regular messages: The messages in the two parts will be sent regularly to each participant. As personalisation is a core process subject to behavioural changes, the content, frequency, and timing of the messages will be determined based on participants' preferences. To save labour and increase efficiency, we will develop a message 'scheduler' program. We will pre-set the message scheduler, which will then automatically send out content to participants according to their preferences. The development of the program is highly useful particularly in cases which participants prefer to receive messages during non-office hours.
   * Therapist-led real-time support messages (chat-type): Chat-based support will be given to the participants as an extension of the regular messages. However, the participants will be informed beforehand that the RA will only play a supportive role and will not provide formal care. The number of the chat messages will not be limited, but the real-time support messages will only be provided during working hours (i.e., 9am-6pm) on weekdays to limit the RA's workload.

Control Group:

The control group will receive instant messages about mental health management from HKSAR Government website (https://www.shallwetalk.hk/en/mental-well-being/mental-well-being-is-related-to-you/), which is open to the public.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged ≥ 50 years; HK-MoCA score range from 18 to 25; MBI-C ≥7; Able to read and communicate in Chinese (Cantonese or Putonghua); Able to use the text or voice messaging function on a smartphone.

Exclusion Criteria:

* Diagnosis of dementia; Diagnosis of psychiatric disease; Currently participating in any type of psychological or behavioural intervention for NPSs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
MBI-C scores | 8 weeks
  The primary outcome will be MBI-C scores to assess NPSs. A higher MBI-C scores will indicate a higher level of neuropsychiatric symptoms.

SECONDARY OUTCOMES:
Depressive symptoms (PHQ-9) | 8 weeks
  Each item was scored on a 4-point scale (0 "not at all" to 3 "nearly every day"). The total score is calculated by summing up the score of all items (range 0-27). High scores indicate worse depressive symptoms.
Anxiety symptoms (GAD-7) | 8 weeks
  A 7-item scale with score ranging from 0 to 21, higher scores indicate higher severity of anxiety symptom
Cognitive functions (HK-MoCA) | 8 weeks
  The total score is calculated by summing up the score of all items. Higher scores indicate better cognitive function.
Acceptance of negative emotions and valued-based actions (AAQ-II) | 8 weeks
  AAQ-II is a measure of psychological flexibility. Each item is rated on a 7-point scale from 1 = never true to 7 = always true. Scores range from 1-49. A lower score indicates a lower level of psychological flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Jae LEE, Principal Investigator — School of nursing, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong